CLINICAL TRIAL: NCT00333996
Title: A Study of the Safety and Efficacy of a New Treatment for Non-Infectious Anterior Uveitis
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 206207-015
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Last update posted 2011-05-30 (Estimated); Status verified 2011-05

CONDITIONS: Anterior Uveitis
MeSH Terms: conditions — Uveitis, Anterior | interventions — Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
This study will evaluate the safety and efficacy of an intravitreal implant of dexamethasone for the treatment of non-infectious anterior uveitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with a diagnosis of non-infectious anterior uveitis in at least one eye

Exclusion Criteria:

* Uncontrolled systemic disease
* Any active ocular infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-05; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Anterior Chamber Cell

CONTACTS AND LOCATIONS:
Overall Officials: Allergan Inc., Study Chair — Allergan
Locations (1):
- Dallas, Texas, United States